CLINICAL TRIAL: NCT02977104
Title: Maestro Handheld Cardiac Monitor Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rakesh Latchamsetty, Assistant Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00074138
Record Dates: First submitted 2016-11-16; First posted 2016-11-30 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: 40 subjects with Atrial Fibrillation 10 subjects with Atrial Flutter 20 subjects with Sinus Rhythm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients in afib or flutter (Other): Maestro ECG
  Interventions: Other: Maestro ECG
- Patients in sinus rhythm (Other): Maestro ECG
  Interventions: Other: Maestro ECG

INTERVENTIONS:
Other: Maestro ECG — Telemetry is obtained through the Maestro handheld ECG device.

SUMMARY:
The purpose of this study is to demonstrate that the Maestro hand held heart monitor can accurately diagnose Atrial Fibrillation, atrial flutter or normal sinus rhythm in patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine if Maestro can be used to detect heart arrhythmias, specifically atrial fibrillation in humans. Maestro will be used to measure heart rate and rhythm at the same time that patients are being monitored with a standard 3, 5, or 12 lead electrocardiogram (ECG) in a clinical setting. The recorded Maestro results will be compared to the ECG results to assess Maestro's accuracy.

Data will be analyzed by a pass/fail criterial. The data will be downloaded and printed for the investigators' interpretation who will first review and code the data from Meastro, blinded to the ECG findings. Then the investigators will interpret the ECG findings and the 2 sets of data will be compared. The ECG result is the true value with which to compare the Maestro result.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide informed consent

Exclusion Criteria:

* implanted pacemakers
* open wounds or abrasions on their hands
* prior damage to hands or thumbs precluding obtaining an ECG tracing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of atrial fibrillation detection | 6 seconds
  Each sample acquired by the Maestro system will be automatically analyzed and rhythm categorized by the automated algorithm. This will then be assessed for accuracy and sensitivity and specificity for detection of atrial fibrillation will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Latchamsetty, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Cardiovascular Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No